CLINICAL TRIAL: NCT03474939
Title: The Effect of Midazolam Premedication on Copeptine Concentration in Blood
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Marek Janiak, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MIDPRECOP
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Preanesthetic Medication; Copeptin
MeSH Terms: conditions — Diabetes Insipidus | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIDAZOLAM (Active Comparator): Patients receive midazolam 7,5mg night before and 60 minutes prior to surgery as part of preanesthetic medication
  Interventions: Drug: Midazolam Oral Tablet
- PLACEBO (Placebo Comparator): Patients receive 1000mg Glucose tablets night before and 60 minutes prior to surgery during premedication
  Interventions: Other: Placebo Oral Tablet

INTERVENTIONS:
Drug: Midazolam Oral Tablet — Midazolam Oral tablet
  Arms: MIDAZOLAM
Other: Placebo Oral Tablet — Glucose 1000mg tablet night before surgery and 60 minutes before surgery
  Arms: PLACEBO

SUMMARY:
The study aim is to assess whether premedication with midazolam prior to surgery affects copeptin concentration in blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery
* Patients with no chronić illness and considered ASA 1 by anesthesiologist
* Patients with mild and controlled chronic illness considered ASA 2 by anesthesiologist

Exclusion Criteria:

* Patient refusal
* Chronic illness requiring intense treatment or uncontrolled illness (ASA 3 or more)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change in copeptin concentration | 48 hours
  Change in the concentration of copeptine measured in blood serum

CONTACTS AND LOCATIONS:
Locations (1):
- I Department of Anesthesiology and Intensive Care Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No